CLINICAL TRIAL: NCT02447614
Title: Follow-up Studies of PS and OSAHS in Chinese Children
Brief Title: Follow-up Studies of Primary Snoring(PS) and Obstructive Sleep Apnea Hypopnea Syndrome(OSAHS) in Chinese Children
Status: Completed | Type: Observational
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Zhifei Xu, The chief of Sleep center, Beijing Children's Hospital
Other Study IDs: BCH-OSAHS-002
Record Dates: First submitted 2015-05-13; First posted 2015-05-19 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: follow up; Primary Snoring; Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Surgery: Adenotonsillectomy
  Interventions: Procedure: Adenotonsillectomy
- Conservative treatment: Mometasone Furoate Aqueous Nasal Spray or uticasone propionate (1/once qd) and（or）Leukotriene antagonists(4 or 5mg/once qn) or H1 receptor antagonists
  Interventions: Other: Conservative treatment
- no treatment: just regular follow-up
  Interventions: Other: no treatment

INTERVENTIONS:
Procedure: Adenotonsillectomy — Adenotonsillectomy
  Groups: Surgery
Other: Conservative treatment — Mometasone Furoate Aqueous Nasal Spray or uticasone propionate (1/once qd) and（or）Leukotriene antagonists(4 or 5mg/once qn) or H1 receptor antagonists
  Groups: Conservative treatment
Other: no treatment — just regular follow-up
  Groups: no treatment

SUMMARY:
The study is designed to investigate the natural course of Primary snoring in 1-2 years or more and the different effect of drug and surgical treatment applied in children with obstructive sleep apnea (OSAS) by comparing the polysomnography(PSG) and sleep questionaires in 6 months after treatment.

DETAILED DESCRIPTION:
The evolution of snoring and OSAS in children is not well established since few studies have been published.This study is designed to evaluate the evolution of primary snoring and OSAS in children who had been submitted to watchful waiting 、drug or adenotonsillectomy.The participated children will be evaluated by full physical examination and nocturnal polysomnography（PSG）, after which they were divided into 2 groups: apnea and snoring. After 6 months following the initial evaluation, patients were submitted to a new nocturnal polysomnography, and all data were compared to those of the first examination.And after 3 months and 12 months following the initial evaluation, patients will be called to complete the sleep questionnaire.Then analyse the change of parameters of polysomnography after 6 months of follow-up,and describe the changes of items of sleep questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-12 yrs, who are referred for clinical evaluation of habitual snoring and who were scheduled for an overnight polysomnogram.

Exclusion Criteria:

* Children who are suffered from any chronic medical or psychiatric condition
* Children with acute respiratory infection
* Children with severe craniofacial deformities
* Children with cardiopulmonary diseases
* Children with a genetic syndrome that was known to affect cognitive abilities, or are receiving medications that are known to interfere with memory or sleep onset or heat rate

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: PS and OSAHS in Chinese children
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
The changes of PSG parameters of children with PS or OSAS | 6 months
  In our study, there are 55 children of mild to moderate SDB with conservative treatment, among which 23 children are chosen in PS group and 32 children are chosen in OSAS group. For PSG, according to the value of OAHI to determine the improvement of the child, the value of OAHI is decreased by ≥ 25% for improvement. In the PS group, there were 2 cases with improvement, and the corresponding remission rate was 8.7%. In the OSAS group, there are 22 cases with improvement, and the corresponding remission rate was 68.8%. There was a significant difference between the remission rate of PS group and that of OSAS group (P<0.001).

SECONDARY OUTCOMES:
The changes of sleep questionnaires of children with PS or OSAS | 3 months, 6 months, 12 months
  There are five impact factors in the PSQ questionnaire, including: 1) nighttime snoring related symptoms (S); 2) sleep accompanying symptoms and related diseases (A); 3) daytime sleepiness related symptoms (L); 4) behavior related symptoms (B); and 5) others' evaluation of children's sleep (O).
  In the PS group, there were significant difference for factor S, A and B at the time of 3 months and one year. For factor L, there was significant change at 3 months, while there was no significant change at half the year and one year.
  In the OSAS group, there was significant change in the S factor for 3 months, half the year, and one year. While for the O factor, there was no significant change in any time. For factor A and L, there was a significant change in 3 months and one year. For the B factor, there was a significant difference at one year.
The changes of level of leukotriene in urine of children with PS or OSAS | 6 months
  There was no significant difference in the level of leukotriene between PS and OSAS group. Also no significant difference in the level of leukotriene was detected among waiting, conservative or surgery group.
The high-sensitivity CRP and Heart rate variability (HRV) of children with SDB | 0 months
  The controls were elder. Children in moderate-severe OSAS group were more boys and more obese. Because of the disease itself, there was statistic difference in AHI, OAI, ODI, respiratoryrelatedarousal index (ArI-resp), average SpO2 and lowest SpO2 among groups.The percentage of high level hs-CRP varied with the severity of SDB and cochran armitage trend test showed statistical significance (Z=-2.5109, p=0.012). In logistic regression analysis, OSAS, otitis media and BMI-z score were independent risk factors for high level hs-CRPafter adjusting for age and gender( p<0.0001). In multiple linear regression,after removing theconfounding factor of OSAS, it showed that high level hs-CRP was negatively correlated with SDNN, RMSSD, LF and HF respectively (p=0.003, p<0.001, p=0.007 and p=0.003 respectively).

OTHER OUTCOMES:
The pictorial memory task acquisition and retention in children with SDB | 0 month
  There was no significant difference in the score of pictorial-based memory task among the control, PS and OSAS groups .Conclusion : Compared with the control group, both PS and OSAS group have abnormal sleep structure and respiratory parameters whereas no significant difference in the score of pictorial-based memory task .We couldn't demonstrate that sleep disordered breathing can affect children's ability of learning picture from the pictorial-based memory task in our study.
The endothelial cell function in children with PS or OSAS | 0 month
  Both mild and moderateesevere OSA groups had lower RHI than PS (P < 0.001, P=0.001, respectively). Linear regression analysis revealed that RHI was positively correlated with age (r=0.17, P=0.002), BMI z score (r=0.14, P=0.008) and oxygen saturation nadir (r=0.15, P=0.006), but negatively correlated with oxygen desaturation index (ODI3%; r=0.19, P=0.001) and respiratory related arousal index (ArI-resp) (r=0.24, P < 0.001). In stepwise regression analysis, age, BMI z score, and ArI-resp were independently associated with endothelial function (r=0.34, P < 0.001).
  Conclusion: Children with OSA are at increased risk for abnormal endothelial function than habitually snoring children. Furthermore, in addition to age and BMI, which are well-established factors affecting endothelial function, both intermittent hypoxia and sleep fragmentation during sleep also emerge as candidate risk factors contributing to endothelial dysfunction in snoring children

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhifei, MD,PhD, Study Director — Beijing Children's Hospital
Locations (1):
- Sleep Center,Beijing Children's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Ward SD, Sheldon SH, Shiffman RN, Lehmann C, Spruyt K; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):e714-55. doi: 10.1542/peds.2012-1672. Epub 2012 Aug 27. PMID 22926176
- [Background] Xu Z, Li B, Shen K. Ambulatory blood pressure monitoring in Chinese children with obstructive sleep apnea/hypopnea syndrome. Pediatr Pulmonol. 2013 Mar;48(3):274-9. doi: 10.1002/ppul.22595. Epub 2012 May 21. PMID 22615200
- [Background] Tan HL, Gozal D, Kheirandish-Gozal L. Obstructive sleep apnea in children: a critical update. Nat Sci Sleep. 2013 Sep 25;5:109-23. doi: 10.2147/NSS.S51907. PMID 24109201
- [Background] Kohler M. Risk factors and treatment for obstructive sleep apnea amongst obese children and adults. Curr Opin Allergy Clin Immunol. 2009 Feb;9(1):4-9. doi: 10.1097/ACI.0b013e32831d8184. PMID 19532087
- [Background] Cheng J, Elden L. Outcomes in children under 12 months of age undergoing adenotonsillectomy for sleep-disordered breathing. Laryngoscope. 2013 Sep;123(9):2281-4. doi: 10.1002/lary.23796. Epub 2013 Jul 2. PMID 23821577
- [Background] Tagaya M, Nakata S, Yasuma F, Mitchell RB, Sasaki F, Miyazaki S, Morinaga M, Otake H, Teranishi M, Nakashima T. Children with severe or moderate obstructive sleep apnoea syndrome show a high incidence of persistence after adenotonsillectomy. Acta Otolaryngol. 2012 Nov;132(11):1208-14. doi: 10.3109/00016489.2012.695088. Epub 2012 Oct 1. PMID 23025449
- [Background] Shen Y, Xu Z, Shen K. Urinary leukotriene E4, obesity, and adenotonsillar hypertrophy in Chinese children with sleep disordered breathing. Sleep. 2011 Aug 1;34(8):1135-041. doi: 10.5665/SLEEP.1178. PMID 21804676
- [Background] Shen Y, Xu Z, Huang Z, Xu J, Qin Q, Shen K. Increased cysteinyl leukotriene concentration and receptor expression in tonsillar tissues of Chinese children with sleep-disordered breathing. Int Immunopharmacol. 2012 Aug;13(4):371-6. doi: 10.1016/j.intimp.2012.05.009. Epub 2012 May 23. PMID 22634478
- [Background] Tapia IE, Marcus CL. Newer treatment modalities for pediatric obstructive sleep apnea. Paediatr Respir Rev. 2013 Sep;14(3):199-203. doi: 10.1016/j.prrv.2012.05.006. Epub 2012 Jun 26. PMID 23931720
- [Background] Friedman BC, Goldman RD. Anti-inflammatory therapy for obstructive sleep apnea in children. Can Fam Physician. 2011 Aug;57(8):891-3. PMID 21841108
- [Background] Kheirandish-Gozal L, Kim J, Goldbart AD, Gozal D. Novel pharmacological approaches for treatment of obstructive sleep apnea in children. Expert Opin Investig Drugs. 2013 Jan;22(1):71-85. doi: 10.1517/13543784.2013.735230. Epub 2012 Nov 5. PMID 23126687
- [Background] Rosen D. Management of obstructive sleep apnea associated with Down syndrome and other craniofacial dysmorphologies. Curr Opin Pulm Med. 2011 Nov;17(6):431-6. doi: 10.1097/MCP.0b013e32834ba9c0. PMID 21918449
- [Background] Heussler H, Chan P, Price AM, Waters K, Davey MJ, Hiscock H. Pharmacological and non-pharmacological management of sleep disturbance in children: an Australian Paediatric Research Network survey. Sleep Med. 2013 Feb;14(2):189-94. doi: 10.1016/j.sleep.2012.09.023. Epub 2012 Dec 12. PMID 23245853
- [Background] Goldbart AD, Greenberg-Dotan S, Tal A. Montelukast for children with obstructive sleep apnea: a double-blind, placebo-controlled study. Pediatrics. 2012 Sep;130(3):e575-80. doi: 10.1542/peds.2012-0310. Epub 2012 Aug 6. PMID 22869829
- [Background] Leboulanger N, Fauroux B. Non-invasive positive-pressure ventilation in children in otolaryngology. Eur Ann Otorhinolaryngol Head Neck Dis. 2013 Apr;130(2):73-7. doi: 10.1016/j.anorl.2012.06.001. Epub 2012 Dec 27. PMID 23273417
- [Derived] Wu Y, Zheng L, Wu P, Tang Y, Xu Z, Ni X. Clinical and PSG Characteristics of Children with Mild OSA and Respiratory Events Terminated Predominantly with Arousal. Can Respir J. 2021 Jun 7;2021:5549423. doi: 10.1155/2021/5549423. eCollection 2021. PMID 34194586
- [Derived] Zhang F, Wu Y, Feng G, Ni X, Xu Z, Gozal D. Polysomnographic correlates of endothelial function in children with obstructive sleep apnea. Sleep Med. 2018 Dec;52:45-50. doi: 10.1016/j.sleep.2018.07.023. Epub 2018 Aug 22. PMID 30269047